CLINICAL TRIAL: NCT01379027
Title: Internet CBT for Depression: Comparing Pure, Guided, and Stepped Care
Brief Title: MoodHelper: Internet Cognitive Behavioral Therapy (CBT) for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH087505 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-06-23 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Depression; Website intervention; CBT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- a treatment as usual (TAU) control condition (No Intervention): Participants will receive recruitment information, go on the study website to enroll and complete assessments over the study web site but will not receive the study intervention.
- Pure self-help Internet CBT for depression (Experimental): Participants will receive TAU plus access to the study website for the self-help Internet CBT for depression, consisting of access to the Internet site without any contact with therapist
  Interventions: Behavioral: Pure self-help Internet CBT for depression
- Guided self-help Internet CBT (Experimental): Participants will receive TAU plus Guided self-help Internet CBT, consisting of access to the Internet site plus brief, periodic telephone contacts with therapists
  Interventions: Behavioral: Guided self-help Internet CBT
- Stepped-Care Internet CBT condition (Experimental): This consists of a Stepped-Care Internet CBT condition, starting with TAU + Pure self-help CBT and progressing to Guided self-help CBT if adequate progress is not observed early on
  Interventions: Behavioral: Stepped-Care Internet CBT condition

INTERVENTIONS:
Behavioral: Pure self-help Internet CBT for depression — Internet, CBT, Depression
  Arms: Pure self-help Internet CBT for depression
Behavioral: Guided self-help Internet CBT — CBT, Depression, Website intervention, coaching
  Arms: Guided self-help Internet CBT
Behavioral: Stepped-Care Internet CBT condition — Depression CBT, Internet intervention
  Arms: Stepped-Care Internet CBT condition

SUMMARY:
Evidence-based treatments (EBTs) for mental health conditions are often not available to persons needing them in the community. Our aim is to test a novel Internet intervention that has the promise of eventually improving the Reach and Implementation of mental health EBTs, speeding the translation of research successes into improved community care.

DETAILED DESCRIPTION:
Evidence-based treatments (EBTs) for depression are often not available to persons needing them; this is particularly true of psychotherapies. Even when available, EBTs are often poorly delivered at less-than-optimal quality. High direct and indirect costs also limit the availability of EBTs. Together these barriers contribute to suboptimal treatment of depression in the community. In a preliminary step toward addressing these quality shortcomings, the investigators propose to conduct a blended efficacy- effectiveness randomized controlled trial (RCT) of high fidelity, Internet-delivered cognitive behavioral therapy (CBT) for depression, extending our previous research to maximize treatment availability and quality as well as to reduce costs. Over a 36-month recruitment period, the investigators will enroll 1,800 adults seeking care for depression from 3 rural healthcare clinics, 3 safety net federally qualified healthcare centers (FQHCs), and 2 non-profit HMOs. Participants will be randomized to: (a) a treatment as usual (TAU) control condition, typically antidepressants and/or psychosocial services; (b) TAU plus Pure self-help Internet CBT for depression, consisting of access to the Internet site without any contact with therapists; (c) TAU plus Guided self-help Internet CBT, consisting of access to the Internet site plus brief, periodic telephone contacts with therapists; or (d) a Stepped-Care Internet CBT condition, starting with TAU + Pure self-help CBT and progressing to Guided self-help CBT if adequate progress is not observed early on. Participants will be followed for one year. The primary hypothesis for which the study is powered is that Guided self-help CBT will result in greater depression symptom improvement than Pure self-help CBT. The investigators also expect secondary analyses to reveal this pattern of results: Guided CBT > Pure CBT > TAU. The investigators will conduct cost-effectiveness analyses (CEA), as the investigators project substantial differences in the direct costs of each study arm. The investigators will also examine TAU healthcare utilization (medications, visits, etc) from electronic medical records (EMR), billing systems, and participant report. The investigators hypothesize that cost per depression free days (DFDs) and quality- adjusted life years (QALYs) will be lowest for Pure CBT, relative to Guided and Stepped-Care CBT and TAU. The investigators also hypothesize that cost per unit of improvement in QALYs and DFDs will be better for Stepped-Care compared to Guided CBT. Additional aims include exploratory examination of secondary outcomes, and predictors and moderators of outcomes among the interventions. The investigators also will collect quantitative and qualitative data on patient, provider, and organizational factors that may impede or facilitate implementation of these interventions, to help prepare for future dissemination efforts. Finally, in this reapplication the investigators have added a non-research Reach Estimation Phase to better estimate acceptance and retention rates under conditions that closely match real-world dissemination

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a score ≥ 10 on the self-report Patient Health Questionnaire (PHQ-8), indicative of clinically significant, moderate depression.
* Participants must identify their primary healthcare provider in one of the 8 performance sites, and give permission to contact him or her for the purpose of periodic progress reports as well as a referral contact in case any emergent crises are detected.
* Participant must be 18 years of age have access to a computer with internet and a working email address.
* Participants must also indicate they are planning to continue receiving services from one of the performance site clinics/organizations for at least the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1816 (Actual)
Dates: Start 2011-10; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The primary hypothesis for which the study is powered is that Guided self-help CBT will result in greater depression symptom improvement than Pure self-help CBT. | assessment measure is administered at baseline and each follow-up, at 5, 10, 15, 25, and 50 weeks after enrollment
  We'll enroll 1,800 adults with depression from 3 rural healthcare clinics, 3 safety net federally qualified healthcare centers and 2 non-profit HMO. Participants will be randomized to: TAU only (b) TAU plus Pure self-help Internet CBT for depression (G-CBT), (c) TAU plus G-CBT, plus brief, periodic therapist telephone contacts; or (d) a Stepped-Care Internet CBT condition, starting with TAU + Pure self-help CBT and progressing to Guided self-help CBT if adequate progress is not observed early on. Participants will be followed for one year.

SECONDARY OUTCOMES:
secondary analyses will examine healthcare utilization for any signs of shifts in amount or mix of TAU services by study condition. | assessment measure is administered at baseline and each follow-up, at 5, 10, 15, 25, and 50 weeks after enrollment
  We will conduct cost-effectiveness analyses, examine TAU healthcare utilization from EMR, participant report and collect quantitative and qualitative data on patient, provider, and organizational factors that may impede or facilitate implementation of these interventions and we have added a non-research Reach Estimation Phase to better estimate acceptance and retention rates under conditions that closely match real-world dissemination

CONTACTS AND LOCATIONS:
Overall Officials: Greg N Clarke, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Sheppler CR, Edelmann AC, Firemark AJ, Sugar CA, Lynch FL, Dickerson JF, Miranda JM, Clarke GN, Asarnow JR. Stepped care for suicide prevention in teens and young adults: Design and methods of a randomized controlled trial. Contemp Clin Trials. 2022 Dec;123:106959. doi: 10.1016/j.cct.2022.106959. Epub 2022 Oct 11. PMID 36228984